CLINICAL TRIAL: NCT00952497
Title: A Phase 2 Open-Label Study Evaluating the Efficacy and Safety of Telatinib in Combination With Chemotherapy as First-Line Therapy in Subjects With Advanced Gastric Cancer
Brief Title: A Study of Telatinib in Combination With Chemotherapy in Subjects With Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ACT Biotech, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEL0805
Record Dates: First submitted 2009-07-30; First posted 2009-08-06 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Gastro-Esophageal Cancer; GE-Junction; Advanced Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cisplatin; Capecitabine; telatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cisplatin, Capecitabine, Telatinib (Experimental)
  Interventions: Drug: Cisplatin, Capecitabine, Telatinib

INTERVENTIONS:
Drug: Cisplatin, Capecitabine, Telatinib — Subjects will receive: Chemotherapy (capecitabine and cisplatin) and telatinib Capecitabine will be administered (1000 mg/m2) twice daily for 14 days followed by a 7-day rest period. Cisplatin (80 mg/m2) will be given as a 1-3 hour infusion once every 3 weeks. Telatinib (3 tablets) will be administered orally, twice daily as a continuous administration. After a maximum of 6 cycles of cisplatin, subjects continue with capecitabine and telatinib or monotherapy with either study drug,depending on the toxicity experienced by the subject, until disease progression.

SUMMARY:
The objectives of this study are to evaluate the anti-tumor activity, safety, and tolerability of telatinib when used in combination with chemotherapy (capecitabine and cisplatin) as first-line therapy in subjects with advanced gastric cancer. The primary objective is to assess progression free survival (PFS) in subjects receiving telatinib in combination with chemotherapy (capecitabine and cisplatin). The secondary objectives are to assess overall survival, overall response rate, safety and tolerability, pharmacokinetics and biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the stomach or gastro-esophageal junction with inoperable locally advanced or metastatic disease, not amenable to curative therapy
* Measurable disease: At least 1 measurable metastatic lesion that has not been irradiated; The lesion will be measured according to RECIST and be evaluated radiologically within 28 days prior to study entry
* ECOG performance status of 0 or 1 at study entry
* Adequate bone marrow, liver and renal function
* Women of childbearing potential:Negative serum pregnancy test within 7 days and must agree to use adequate contraception (barrier method of birth control) prior to study entry, for the duration of study participation and 28 days after the last study drug dosing

Exclusion Criteria:

* Previous chemotherapy for locally advanced or metastatic gastric cancer:prior neoadjuvant or adjuvant chemotherapy completed at least 6 months prior to study entry is allowed
* Previous anti-angiogenic therapy: Anti VEGF or VEGFR tyrosine kinase inhibitor such as bevacizumab, sorafenib, sunitinib, AZD2171
* Previous total platinum dose >300 mg/m2: total prior platinum dose of ≤300 mg/m2 will be allowed in the adjuvant or neo-adjuvant setting
* Candidates for curative therapy
* Clinical or radiographic evidence of brain metastasis
* Cardiac disease; uncontrolled hypertension; hemorrhage/bleeding events
* Known or suspected allergy to any component of telatinib, cisplatin or capecitabine
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Unable to take oral medications that could affect oral intake of capecitabine and telatinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The primary objective is to assess progression free survival (PFS). PFS will be measured from the date of first study drug administration to the date of first scan that first documents disease progression. | 6 months

SECONDARY OUTCOMES:
Other efficacy variables are overall survival, overall response rate, safety and tolerability. Exploratory analyses may be performed to investigate the correlation of biomarker status with treatment effect and response. | 18 months from start of enrollment to evaluation of primary endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Scott Freeman, MD, Study Director — ACT Biotech, Inc
Locations (11):
- United States (5):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Central Georgia Cancer Care, P.C., Macon, Georgia
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - The West Clinic, Memphis, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Spain (6):
  - Hospital Vall d' Hebron, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander